CLINICAL TRIAL: NCT03060915
Title: Comparison of Actigraphy Sleep Parameters vs Polysomnography Sleep Parameters in OSA Patient's
Brief Title: Actigraphy Sleep Parameters in Obstructive Sleep Apnea Patient's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Montserrat, Medical doctor, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACT_2017
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Actigraphy; Polysomnography; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography; Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polysomnography and actigraphy (Other): Polysomnography and actigraphy
  Interventions: Device: Polysomnography; Device: Actigraphy

INTERVENTIONS:
Device: Polysomnography — Patient's undergo a polysomnography
Device: Actigraphy — Patient's wear an actigraphy while doing the polysomnography

SUMMARY:
Those patient's that come to the sleep unit and that accept to participate in the study will undergo a polysomnography with the extra of an actigraphy placed in their no dominant arm wrist. The outcomes that will be analyzed are:

Time in bed, assumed sleep time, wake time, sleep efficiency, sleep latency, light's on/light's off

ELIGIBILITY:
Inclusion Criteria:

* Patient's with OSA suspicion undergoing a PSG in the sleep unit

Exclusion Criteria:

* Neurologic disorders
* Severe comorbidities
* Other sleep disorders, such as insomnia
* No informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Sleep time (min) | 3 months
  To compare the outcomes acquired with the actigraphy with those acquired by the Polysomnography

SECONDARY OUTCOMES:
sleep efficiency | 3 months
  To evaluate the agreement, sensitivity and specificity between the outcomes acquired by the Polysomnography and by the actigraphy.
Wake time | 3 months
  To evaluate the agreement, sensitivity and specificity between the outcomes acquired by the Polysomnography and by the actigraphy.
sleep latency | 3 months
  To evaluate the agreement, sensitivity and specificity between the outcomes acquired by the Polysomnography and by the actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Montserrat, MD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No